CLINICAL TRIAL: NCT02496572
Title: Effectiveness of a Simplified Short Regimen for Multidrug Resistant Tuberculosis Treatment in Karakalpakstan, Uzbekistan
Brief Title: Effectiveness of a Simplified Short Regimen for Multidrug Resistant Tuberculosis in Uzbekistan
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medecins Sans Frontieres, Netherlands (Other)
Collaborators: Ministry of Health, Republic of Uzbekistan (Other Government); Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: MSF MDRTB Uzbek
Record Dates: First submitted 2014-07-02; First posted 2015-07-14 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Multidrug Resistant Tuberculosis
Keywords: Tuberculosis, multidrug resistant; Short-course regimen; Medecins sans Frontieres, MSF; Uzbekistan, Ministry of Health
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Jacobs syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Short-course MDR-TB regimen patients: Short course MDR-TB treatment regimen. New presumptively diagnosed MDR TB patients (adults and children) with Xpert® MTB/RIF or Hain MTBDR, or confirmed with Hain MTBDR plus on positive cultures if initial molecular tests negative or confirmed from MGIT culture/DST if initial molecular tests negative;
  Children (<14 years old) suspected of MDR TB without bacteriological confirmation but documented as a close contact of a confirmed MDR TB patient
  Interventions: Drug: Short course MDR-TB treatment regimen

INTERVENTIONS:
Drug: Short course MDR-TB treatment regimen — Intensive phase:
  Pyrazinamide (Z) + Ethambutol (E) + Isoniazid (H) + Moxifloxacin (Mfx) + Capreomycin (Cm) + Prothionamide (Pto) + Clofazimine (Cfz) for at least 4 months and until one negative culture is documented with a maximum of 6 months duration.
  Continuation phase:
  Continuation phase of Pyrazinamide (Z) + Ethambutol (E) + Moxifloxacin (Mfx) + Prothionamide (Pto) + Clofazimine (Cfz) for fixed 5 months duration.
  Other Names: Bangladesh protocol; Shortened course MDR-TB treatment; 9-month MDR-TB regimen

SUMMARY:
Multidrug resistant tuberculosis (MDR TB) is a growing problem and few people have access to adequate diagnosis and treatment. The current recommended treatment regimen for MDR TB has a minimum of 20 months duration with high toxicity. Scale up of MDR TB treatment is associated with high default rates, and experience in the Medecins Sans Frontieres (MSF) programme in Uzbekistan shows that the current standard treatment greatly limits the ability to scale up to meet the high rates of MDR TB in the region.

Evidence from Bangladesh in 2010 showed that a 9-month short-course regimen could achieve a relapse-free cure rate of 88%. Several countries in West Africa started implementing similar regimens with similar outcomes. Evidence of effectiveness of this shortened regimen among regions with high second line drug use and resistance is still limited.

The investigators propose an observational study under programmatic conditions to evaluate the effectiveness of a shortened course MDR TB regimen in the high MDR/extensively drug resistant (XDR) TB prevalence and high second-line drug resistance setting of Karakalpakstan, Uzbekistan.

DETAILED DESCRIPTION:
A prospective observational study has been designed. The study regimen is composed of an intensive phase of at least 4 months duration of Pyrazinamide (Z) + Ethambutol (E) + Isoniazid (H) + Moxifloxacin (Mfx) + Capreomycin (or Kanamycin/Amikacin) (Cm/Km/Am) + Prothionamide (Pto) + Clofazimine (Cfz) and a continuation phase of oral drugs Z-E-Mfx-Pto-Cfz. Patients will be followed up until the end of treatment and during 12 months after treatment completion in order to evaluate the rate of relapse.

Data will be recorded in patient's clinical files and electronic databases and analyzed with Stata 11.0.

This study is a result of ongoing collaboration of MSF with the Ministry of Health in Uzbekistan; results will be shared with the national health authorities, World Health Organization and the rest of the scientific community and aim to influence and improve treatment and care of patients with MDR TB.

ELIGIBILITY:
Inclusion Criteria:

* New presumptively diagnosed MDR TB patients (adults and children) with Xpert® MTB/RIF (rifampicin) or Hain MTBDR (Mycobacterium tuberculosis drug resistance), or confirmed with Hain MTBDR plus on positive cultures if initial molecular tests negative or confirmed from MGIT (mycobacteria growth indicator tube) culture/DST if initial molecular tests negative;
* Children (<14 yo) suspected of MDR TB without bacteriological confirmation but documented as a close contact of a confirmed MDR TB patient; AND
* Informed consent to participate in the study signed by the patient or the responsible caretaker for patients <16 years old (as per national legislation).

Only patients with a history of prior treatment with second line anti-TB drugs for less than one month will be eligible for inclusion.

Patients will be included regardless of HIV status.

Exclusion Criteria:

* Baseline contraindications to any medications of the study regimen medications, where benefits of the regimen do not outweigh the risks as judged by treating physician;
* Severe renal insufficiency with estimated creatinine clearance of <30 ml/min at baseline (calculated with Cockcroft-Gault formula);
* Patients with extrapulmonary TB only (without involvement of lung parenchyma)
* Patients with documented ofloxacin resistance
* Patients with XDR TB (additional resistance to SLD [second line drug] kanamycin (or capreomycin) AND ofloxacin);
* Patients with resistance to both Km and Cm.
* Critically ill and in the judgement of the treating physician unlikely to survive more than 1 week (these patients may still be commenced on standard MDR TB treatment according to the Karakalpakstan comprehensive TB treatment guidelines)
* Has one or more of the following risk factors for QTc prolongation:
* A confirmed prolongation of QTc interval (Fridericia formula), e.g., repeated demonstration of QTcF (Fridericia correction) interval > 500 ms in the screening ECG (i.e., retesting to reassess eligibility will be allowed once using an unscheduled visit during the screening phase)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be referred from the facilities described below in three districts in Karakalpakstan, Uzbekistan
  1. Kegeily Rayon: Kegeily rayon is a large rayon (district) with a population of 83,000. The rayon has 2 Polyclinics (outpatient clinics for TB care) and 21 SVPs (general practice surgeries with staff trained in TB care).
  2. Shumanay Rayon. A small rayon close to Khodjeily rayon with a population of 52,000. There is 1 Polyclinic and 9 SVPs in the rayon
  3. Nukus City Nukus city is the largest district in Karakalpakstan with a population of 268 000. There are 9 polyclinics.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-03 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Rate of relapse-free success at 12 months follow-up (composite measure of the percentage of patients obtaining cure and treatment completion) | End of treatment to 1 year following completion of a 9-11 month treatment regimen

SECONDARY OUTCOMES:
Predictive value of 1st and 2nd line drug resistance at baseline on treatment outcomes (proportion classified as sensitive amongst ethambutol, pyrazinamide, capreomycin and kanamycin) | 1 year following completion of a 9-11 month treatment regimen
Rate of adverse events (proportion of patients experiencing at least one adverse event) | 1 year following completion of a 9-11 month treatment regimen
Rate of treatment interruptions (proportion of patients missing treatment >1 day of complete regimen) | At completion of 9-11 months treatment regimen
Rate of unfavorable outcomes whilst on treatment (composite of patients with default, death, failure) during study period | At completion of 9-11 months treatment regimen
Agreement between smear microscopy and culture (expressed as a kappa coefficient) | At completion of 9-11 months treatment regimen
Proportion of patients with amplification in drug resistance (defined as a patient previously testing sensitive to a drug who subsequently tests resistant) on follow-up drug susceptibility testing compared with baseline. | 1 year after completion of 9-11 months treatment regimen
Rate of treatment modifications (composite measure of proportion of patients requiring cessation or replacement of a drug due to adverse events not described in the protocol) | At completion of 9-11 months treatment regimen
Rate of successful outcomes at end of treatment (composite of patients with treatment outcomes cured and completed ) | At completion of 9-11 months treatment regimen
Rate of adverse events by organ group (categorised as cardiac, respiratory, gastrointestinal, auditory, systemic, dermatological, opthalmologic, neurological, other) | 1 year after completion of 9-11 months treatment regimen
Severity of adverse events (proportion of adverse events classified as mild, moderate, severe and potentially life-threatening) as per DAID criteria | 1 year after completion of 9-11 months treatment regimen
Number of missed days in patients missing >1 day of treatment | At completion of 9-11 months treatment regimen

CONTACTS AND LOCATIONS:
Overall Officials: Philipp du Cros, MBBS, Principal Investigator — Medecins sans Frontieres (MSF); Khamraev A Karimovich, MD, Principal Investigator — Ministry of Health, Republic of Uzbekistan
Locations (1):
- Outpatient clinics in three districts, Nukus, Karakalpakstan, Uzbekistan